CLINICAL TRIAL: NCT05860283
Title: Core Stability Exercise Versus Diaphragmatic Release on Respiratory Functions on Physical Therapists With Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sumaya Serageldin Mohamed, Physical therapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Respiratory functions in LBP
Record Dates: First submitted 2023-03-18; First posted 2023-05-16 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Mechanical Low Back Pain; Respiratory Functions
Keywords: Core stability exercises; Diaphragmatic release technique
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Core stabilization exercise group (Active Comparator): Core muscle activation exercises will be done using the pressure biofeedback unit. The session will include visual, auditory & tactile biofeedback. Visual monitoring of the pressure gauge by the subjects during the exercise will be allowed and breath holding or compensatory movements will be avoided.
  Interventions: Device: Core stabilization exercise using pressure biofeedback unit
- Diaphragmatic release group (Active Comparator): The subjects will lay supine with relaxed limbs. Positioned at the head of the subjects, there will be manual contact with the pisiform, hypothenar region and the last three fingers bilaterally to the underside of the seventh to tenth rib costal cartilages, with the forearms aligned toward the subject's shoulders. In the inspiratory phase, a gentle pull will be given at the points of contact with both hands in the direction of the head and slightly laterally, accompanying the elevation of the ribs. During exhalation, a deepened contact will be given towards the inner costal margin, to resist the rebounding movement of the thoracic cage. In the subsequent respiratory cycles, there will be a progressive increase in the depth of contact inside the costal margin.
  Interventions: Procedure: Diaphragmatic release technique
- Control group (No Intervention): The subjects in this group will receive traditional physical therapy program only.

INTERVENTIONS:
Device: Core stabilization exercise using pressure biofeedback unit — From crook lying:
  * 1st and 2nd weeks LEVEL 1: ADIM and hold for 10 seconds LEVEL 2 : Hold for 5 sec. Repeat 10 times. Opposite lower extremity on plinth; bent leg fall out.
  * 3rd and 4th week LEVEL 3 : Opposite lower extremity on plinth a)Lift bend leg to 90˚ hip flexion b)Slide heel to extend knee c)Lift straight leg to 45˚.
  * 5th and 6th weeks LEVEL 4 : Hold opposite lower extremity at 90˚ of hip flexion a)Lift bend leg to 90˚ hip flexion b)Slide heel to extend knee c)Lift straight leg to 45˚.
  From prone lying:
  Extension of each lower extremity. The exercise progression each week will be evaluated.Each exercise session lasted 20 min. The patients had to hold each exercise for 10 seconds, three sets per session and each set 10 repetitions.
  Arms: Core stabilization exercise group
Procedure: Diaphragmatic release technique — This technique will be given 3 days per week for 6 weeks with total technique duration of 45 minutes. The maneuver will be repeated in 4 sets per session, each set will consist of 5 deep breaths with 2-min intervals in between sets.
  Arms: Diaphragmatic release group

SUMMARY:
To compare between core stability exercise and diaphragmatic release on respiratory functions on physical therapists with low back pain.

DETAILED DESCRIPTION:
Low back pain is the most frequent self-reported type of musculoskeletal pain. It is often recurrent and has important socioeconomic consequences. 99.5% of Egyptian physical therapists (PTs) suffer from work related musculoskeletal disorders (WMSDs), mainly in the lower back (69.1%) and it is more common in female than male therapists. Physical therapists are routinely exposed to work-related physically demanding tasks such as handling heavy patients, applying manual techniques and assuming sustained awkward positions, which are the most common predisposing factors for development of WMSDs.

Respiratory dysfunction is a major factor for the diagnosis and treatment of chronic LBP. This respiratory dysfunction may be related to the altered function of the diaphragm and poor coordination of deep stabilization muscles due to dysfunctional movement patterns. Respiratory dysfunction compromises the subject's ability to stabilize the spine during balancing and postural tasks. Besides diaphragmatic dysfunction, several studies have observed in chronic LBP delayed or decreased activation of lumbar multifidi and transversus abdominus during gait and extremity movement. Since it is difficult to isolate contraction of the transversus abdominis required for the core stability exercises, biofeedback strategies using pressure biofeedback unit (PBU) will be used. This instrument allows visual detection of pressure fluctuations inherent to movements in that region. Another clinical use for the PBU is to help train lumbopelvic stability in individuals with chronic LBP during open-chain segmental control exercises, through challenging the motor control by active movements of the upper or lower limbs, meanwhile the individuals should maintain lumbopelvic neutral position known by getting visual feedback of maintenance of a steady pressure.

People with LBP have an abnormal diaphragm position impacted by small diaphragmatic excursions (mobility) with respiration, in other words "the diaphragm is splinted". Diaphragm tightness can promote shallow breathing, resulting in decreased diaphragm contractile force that impacts the diaphragm strength. Diaphragmatic release has an immediate effect on the diaphragm strength. Increased diaphragm strength immediately follows the intervention, suggesting utility of these techniques for patients with diaphragmatic movement restrictions or breathing-related disorders.

By reviewing the literature it was found that both core stability exercises and diaphragmatic release techniques have positive effects on both respiratory variables & low back pain. Thus, the present study will compare between these two interventions.

ELIGIBILITY:
Inclusion criteria:

* Female physical therapists from 25 to 35 years of age.
* Body mass index less than 30.
* Mechanical LBP persisting for at least 6 months upto1 year with at least three episodes of LBP symptoms for the previous six months.
* Pain score range between 3 and 7 on the Numerical Pain Rating Scale (NPRS) and able to perform the experiment procedure without symptom aggravation.
* Oswestry disability index (ODI) of 7 or higher.
* Did not participate regularly in any training program or manual therapy intervention during the last 6 months.

Exclusion criteria:-

* Current and former smokers.
* Body mass index of 30 or higher.
* Numerical pain rating scale higher than 7 as they will not be able to perform maximum contraction.
* Participants with a history of acute traumatic low back pain in previous two months.
* Lumbar, abdominal, or gynaecological surgery in the past year ,disc herniation or spinal fracture; irradiated pain to the leg; neurological , respiratory and cardiovascular pathologies and infectious health problems.
* Menstruating women, pregnancy or postpartum.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — participant eligibility is based on self-representation of gender identity
Enrollment: 90 (Estimated)
Dates: Start 2023-07-04 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Pulmonary Function tests | one year
  Test will be performed with a spirometer device. Forced vital capacity (FVC) in litres, forced expiratory volume in 1st second (FEV1) in litres, the ratio between FEV1/FVC in litres, peak expiratory flow rate (PEFR) in litres/min and minute volume ventilation (MVV) in litres/min will be measured by spirometer
The diaphragm excursion and thickness | one year
  They will be assessed with ultrasound M-mode and B-modes, respectively.Diaphragm excursion ( in cm) will be taken during both quiet breathing (QB) and deep breathing (DB). The diaphragm thickness (in mm) will be measured at the end of inspiration (Tins) and expiration (Texp) during DB. Diaphragm thickness change is calculated by this formula: (Tins _ Texp)/Texp *100.
Total Faulty Breathing Scale (TFBS) | one year
  Total faulty breathing scale will be used to assess faulty breathing pattern during quiet and deep breathing in an upright standing position. The presence or absence of faulty breathing is the outcome variable, to be assessed by observation of lifting of the clavicle, lateral rib motion, and abdominal movement which will be categorized on a scale of normal (0), mild (1-4), moderate (5-8), and severe (9-12). Higher scores indicate a worse outcome.
Chest expansion | one year
  It will be measured (in cm) using a tape measure. The three positions for measurement will be: 1) the upper chest, under the armpit mid-sternal line; 2) the lower chest, the xiphoid process mid-sternal line; and 3) the abdomen, at the umbilical area.

SECONDARY OUTCOMES:
Numerical pain rating scale (NPRS) | one year
  Numerical pain rating scale is for rating pain intensity. Subjects will be asked to score the pain intensity over the last 24 hours on the NPRS. The scale range between 0 and 10, with 0 being no pain and 10 being worst pain.
Oswestry Disability Index (ODI) | one year
  Oswestry disability index is a clinical assessment tool that will provide an estimate of LBP disability expressed as a percentage score.It consists of ten sections or items to assess pain, personal care, lifting, walking, sitting, standing, sleeping, sex life (if applicable), social life and travelling. Each item is scaled from 0 to 5. The rating is: "Patient Score = (Patient's score/Possible maximum score) × 100". A score of 0% means minimal disability, and a score of 100% means bed addiction. High scores in this scale indicate worse outcomes.
Pressure biofeedback unit (PBU) | one year
  A three-chamber air-filled pressure cell, a catheter and a sphygmomanometer gauge used to assess core stability (in mmHg). The subjects will perform the Sahrmann five level core stability test. The starting pressure during this test is 40 mmHg and the subjects should be able to maintain this pressure in all the 5 levels of the test while performing abdominal drawing in maneuver for 10 seconds. Compensatory postures (holding of breath, movement of the pelvis, visible, or evident contraction of the External oblique muscle, and pressing of the heels toward the floor) indicates weak core muscles.

CONTACTS AND LOCATIONS:
Overall Officials: Alaa El-Moatasem, Doctoral, Study Director — Departement of Cardiovascular Respiratory Disorder and Geriatrics- Faculty of Physical Therapy- Cairo University; Rehab ElSawy, doctoral, Study Director — Chest Diseases Departement - Faculty of Medicine - Benha University
Locations (1):
- Faculty of physical therapy- Cairo University, Cairo, Egypt